CLINICAL TRIAL: NCT01267773
Title: Treatment of Youth Comorbid Conduct Problems and Depression
Brief Title: Treatment of Conduct Problems and Depression
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Jennifer Wolff, Staff Psychologist, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH086606
Record Dates: First submitted 2010-11-16; First posted 2010-12-29 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Depression; Oppositional Defiant Disorder; Conduct Disorder
Keywords: depression; conduct problems
MeSH Terms: conditions — Depression; Oppositional Defiant Disorder; Conduct Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential Treatment (Active Comparator)
  Interventions: Behavioral: Integrated Treatment
- Integrated Treatment (Experimental)
  Interventions: Behavioral: Integrated Treatment

INTERVENTIONS:
Behavioral: Integrated Treatment

SUMMARY:
Having both depression and conduct problems at the same time has been found to be associated with increased risk for the other and increased risk of negative outcomes. This study will develop an family based cognitive behavioral treatment protocol for youths with both conduct problems and depression, that will take be administered over the course of six months. Youth with comorbid conduct problems and depression will be assigned to the experimental condition or treatment as usual in a community care setting. The treatment manual will be revised as needed. Youth will be assessed before and after treatment to examine program potential. The goal of this research is to develop a more comprehensive outpatient treatment for youth with both conduct problems and depression.

ELIGIBILITY:
Inclusion Criteria:

* 8-14 years old
* Diagnosis of ODD or CD
* Diagnosis of Depression
* Speaks English

Exclusion Criteria:

* Developmental/cognitive delays
* Substance dependence
* Psychotic disorder or symptoms

Ages: 8 Years to 14 Years | Sex: All
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Depression Symptoms | baseline to week 24
  Change in depression symptoms from baseline to week 24 will be measured using the Children's Depression Inventory
oppositional symptoms | baseline to week 24
  change in symptoms of oppositionality from baseline to week 24 will be measured using the Disruptive Behavior Disorders Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Wolff, PhD, Principal Investigator — Rhode Island Hospital/Brown University; Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States